CLINICAL TRIAL: NCT01984970
Title: Evaluation McGrath Series 5 Videolaryngoscope for Double-lumen Tube Intubation
Brief Title: McGrath Series 5 Videolaryngoscope for Double-lumen Tube Intubation
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, M.D., Ph.D., Attending physician, Huazhong University of Science and Technology
Other Study IDs: 20121126001
Record Dates: First submitted 2013-11-01; First posted 2013-11-15 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Intubation; Difficult; Intubation Complication
Keywords: McGrath Videolaryngoscope; double-lumen tube intubation; Thoracic surgery

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- videolaryngoscope: The patients received videolaryngoscope for double-lumen tube intubation
  Interventions: Device: videolaryngoscope

INTERVENTIONS:
Device: videolaryngoscope — McGrath Series 5 videolaryngoscope is one kind of portable videolaryngoscopes, which has been usde in both unexpected and anticipated difficult intubation.

SUMMARY:
1. Double-lumen tube intubation is difficult, compared with single lume tube.
2. McGrath Series 5 videolaryngoscope hase been used in difficult airway management, both in anesthetized and awake patients.
3. But there was little information about McGrath Series 5 videolaryngoscope for double-lumen tube intubation.

DETAILED DESCRIPTION:
In this study, the purpose was to evaluate the success rate and intubation time of McGrath Series 5 videolaryngoscope for double-lumen tube intubation in patients without predictors of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* thoracic surgery
* ASA classification 1-3

Exclusion Criteria:

* Emergent operation
* predicted difficult airway
* difficult ventilation
* limited mouth opening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients scheduled for thoracic surgery requiring double-lumen tube insertion for one-lung ventilation
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
intubation time | at intubation
  defined as time from inserting blade to mouth to three cycles on capnograph

SECONDARY OUTCOMES:
number of successful intubation at first attempt | at intubation

OTHER OUTCOMES:
BMI | one day before operation
mouth opening | one day before operation
  measure with a ruler
Thyromental distance | one day before operation
  measure with a ruler
Airway evaluation with Mallampati Score | one day before operation
  based on the modified Mallampati classification. degree 1 to 4
Airway evalutaion with Cormack-Lehane Score | at intubation
  based on Cormack-Lehane classification. degree 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, Ph.D.,M.D., Study Director — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Yao WL, Wang XR, Xu H, Zhang Y, Zhang CH. McGrath((R)) series 5 videolaryngoscope evaluation for double-lumen tube intubation. Anaesthesia. 2014 Jun;69(6):646-7. doi: 10.1111/anae.12720. No abstract available. PMID 24813140